CLINICAL TRIAL: NCT06767930
Title: Effects of Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) in Adults with Bilateral Cerebral Palsy
Brief Title: Effects of HABIT-ILE in Adults with Bilateral Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Paris 12 Val de Marne University (Other)
Responsible Party: Principal Investigator, Yannick Bleyenheuft, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B403201316810i
Record Dates: First submitted 2025-01-05; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy; Bilateral Cerebral Palsy
Keywords: cerebral palsy; motor skill learning; intensive therapy; body function; body structure; muscle structure; pain; activities; quality of life; adults
MeSH Terms: conditions — Cerebral Palsy; Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: The trial will be a single-blind, randomized controlled trial. Participants will be randomly assigned to one of two groups: a control group receiving conventional therapy or a treatment group participating in the HABIT-ILE therapy program. Longitudinal assessments will be conducted the week before the intervention, at the end of the two-week intervention and three months post-intervention.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HABIT-ILE (Experimental)
  Interventions: Behavioral: Hand and Arm Bimanual Intensive Therapy Including Lower Extremities
- Conventional intervention (Active Comparator)
  Interventions: Behavioral: Conventional intervention

INTERVENTIONS:
Behavioral: Hand and Arm Bimanual Intensive Therapy Including Lower Extremities — The HABIT-ILE (Hand-Arm Bimanual Intensive Therapy Including Lower Extremities) program is an intensive rehabilitation therapy designed to improve motor functions and promote functional independence. Participants in this arm will engage in 6.5 hours of structured activities per day for two weeks (10 days). The therapy focuses on bimanual coordination combined with constant stimulation of the trunk and/or lower extremities, using task-oriented exercises tailored to individual goals. Each participant will be supported by one or two therapists and supervised by a trained team to ensure the program is delivered effectively and safely. The therapy emphasizes engaging, play-based activities to maximize motivation and active participation.
  Arms: HABIT-ILE
Behavioral: Conventional intervention — Participants in the control group will continue their usual care, which includes conventional physical and occupational therapy, for a duration of two weeks. They will follow their regular therapy schedules without any changes to their routines or treatment habits. This approach ensures that the control group reflects standard rehabilitation practices, allowing for a direct comparison with the intervention group.
  Arms: Conventional intervention

SUMMARY:
This randomized controlled trial (RCT) aims to evaluate the effects of intensive Hand and Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) in improving body structure, function, daily activities, and participation outcomes among adults with cerebral palsy.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will investigate the impact of two weeks of HABIT-ILE therapy versus conventional rehabilitation on spinal, muscular, and functional outcomes in adults (18-50 years old) with bilateral cerebral palsy (CP). Key assessments will include changes in gross motor function, spinal and muscular adaptations assessed via EMG and ultrasound, strength testing, clinical motor function tests, pain assessment, and questionnaires on activity and participation. This study aims to provide a comprehensive analysis of HABIT-ILE's effects especially on motor function, daily life activities and participation across a wide range of age.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed bilateral cerebral palsy,
* Adults aged 18 to 50 years old,
* Level of manual ability : level I to V of MACS
* Level of gross motor function : level I to IV of GMFCS
* Ability to follow instructions and complete testing,
* Ability to walk 10 meters independently without human assistance (technical aids such as orthoses or walking aids are permitted).

Exclusion Criteria:

* Unstable seizure
* Programmed botulinum toxin or orthopedic surgery in the 6 months before the intervention, during intervention period or 6 months after the intervention time
* Alcohol/drug abuse
* Pregnancy
* Severe visual or cognitive (severe aphasia, psychiatric conditions) impairments likely to interfere with intervention or testing session completion
* Uncontrolled health issues (cardiac, metabolic...)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Gross Motor Function Measurement (GMFM-66) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Measurement of change in gross motor function over time in adults with cerebral palsy.

SECONDARY OUTCOMES:
Changes in muscle strength (Biodex System 4 pro®) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Measurement of maximal isometric muscle strength for specific lower limb and upper limb muscles using a Biodex System 4 pro® (Biodex Medical Systems, Inc., Shirley, NY, USA) isokinetic device.
Changes in muscle strength (Jamar) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Measurement of grip strength using the Jamar dynamometer.
Changes in muscle range of motion (Biodex System 4 pro®) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Assessment of passive and active range of motion for targeted joints using the Biodex System 4 Pro® dynamometer (Biodex Medical Systems, Inc., Shirley, NY, USA).
Changes in neuromuscular command (muscle co-contraction) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Evaluation of muscles co-contraction in lower limbs and upper limbs by combining isometric force measurements with electromyography (EMG) recordings to monitor the activation patterns of agonist and antagonist muscles during contractions.
Changes in unimanual dexterity (Box and Blocks Test - BBT) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Measurement of gross manual dexterity by counting how many blocks a participant can transfer from one side of a box to the other in one minute
Changes in the 2-Minutes' Walk Test (2MWT) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Measurement of the maximum distance covered by the patient in a 2-minutes' walk test, assessing the endurance and walking ability over a short duration.
Changes in spinal function (electromyography - EMG) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Evaluation of spinal function through electromyography (EMG) during the 2-minutes' walk test, assessing muscle activation and coordination of the spinal cord during walking
Changes in pain perception (Quantitative Sensory Testing - QST) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Measurement of sensory response to determine pain threshold and pain perception.
Changes in daily pain perception (Ecological Moment Assessment) | Pre-intervention (1 week before), during intervention (camp or control period), post-intervention (1 week after), 3 months follow-up
  Ecological assessment of daily pain perception using a smartphone application sending randomized notifications throughout the day to prompt the patient to report their pain levels.
Changes in severity of pain (Brief Pain Inventory - Short Form - BPI-SF) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing the severity of pain and its impact on functioning.
Changes in neuropathic pain (PROMIS PQ-Neuro) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire designed to identify patients likely experiencing neuropathic pain and to assess its severity.
Changes in perception of pain (Pain Catastrophizing Scale - PCS) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing the extent of catastrophic thinking related to pain, including rumination, magnification, and helplessness, across three subscales. The total score ranges from 0 to 52 (higher scores indicate a greater degree of pain catastrophizing).
Changes in coping strategies (Coping Strategies Questionnaire - CSQ-F) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing five cognitive coping strategies for managing pain-distraction (attention diversion), catastrophising, praying and hoping, ignoring pain sensations, and reinterpreting pain sensations-based on the frequency of use for each strategy.
Changes in coping strategies (General Self-Efficacy Scale - GSES) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing the belief in one's ability to handle various difficult situations. Scores range from 10 to 40 (lower scores suggest reduced self-efficacy).
Changes in daily activities (Canadian Occupational Performance Measure - COPM) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  The COPM measures the patient's self-perception of occupational performance and satisfaction of it in daily activities over time. It ranges from 1 to 10, a higher score means a better performance.
Changes in daily activities (ABILHAND Questionnaire) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing the patient's performance in unimanual and bimanual upper limb activities, with scores ranging from -6 to +6 logits (higher score indicates better performance).
Changes in daily activities (ACTIVLIM-CP Questionnaire) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing the patient's ability to perform daily activities using the upper and/or lower limbs, with scores ranging from -5 to +5 logits (higher scores indicates better performance).
Changes in daily activities (ABILOCO questionnaire) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing the patient's ability to perform daily activities using the lower limbs, with scores ranging from -4 to +4 logits (higher scores indicates better performance)
Changes in participation (Participation in Life Situation Questionnaire - PILS) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing the participation and engagement in life situation, assessing how cerebral palsy affects the patient's ability to participate in various activities and social situations.
Changes in psychological well-being (Hospital Anxiety and Depression Scale - HADS) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing the patient's level of anxiety and depression, with scores ranging from 0 to 21 for both subscales (higher scores indicate higher levels of anxiety of depression).
Changes in pain and sleeping (Pain and Sleep Questionnaire 3 - PSQ-3) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing the impact of pain on sleep quality. Scores range from 0 to 30 (higher scores indicate greater disruption to sleep due to pain).
Changes in fatigue (Multidimensional Fatigue Inventory - MFI) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing fatigue across five dimensions: general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation. Each subscale score ranges from 4 to 20 (higher scores indicate more severe fatigue in the respective domain).
Changes in quality of life (WHOQOL-BREF) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing quality of life across four domains: physical health, psychological health, social relationships, and environment. Scores for each domain range from 4 to 20 (higher scores indicate better quality of life).
Changes in cognitive function (PROMIS Neuro-QOL Short Form Cognitive Function 2.0) | pre-intervention (1 week before), post-intervention (1 week after), 3 months follow-up
  Questionnaire assessing perceived cognitive function, focusing on areas such as memory, attention, and problem-solving. It is a 4-item questionnaire, each item uses a 5-point Likert scale ranging from 1 ("Never") to 5 ("Always"), with higher scores indicating worse cognitive functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculté des Sciences de la Motricité (UCLouvain), Louvain-la-Neuve, Brabant-Wallon, Belgium

IPD SHARING:
Plan to Share IPD: No